CLINICAL TRIAL: NCT02421666
Title: A Comparative Trial of Improving Care for Underserved Asian Americans Infected With HBV
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Temple University (Other)
Collaborators: Patient-Centered Outcomes Research Institute (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Supportive Care
Other Study IDs: PCORI-HBV
Record Dates: First submitted 2015-04-10; First posted 2015-04-21 (Estimated); Results first posted 2020-10-08 (Actual); Last update posted 2020-10-08 (Actual); Status verified 2020-10

CONDITIONS: Hepatitis B
MeSH Terms: conditions — Hepatitis B

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- behavioral PNMI (Experimental): eligible patients received patient navigator led plus mobile phone text messaging intervention(PNMI) or standard care.
  Interventions: Behavioral: PNMI
- control (No Intervention): eligible chronic HBV patients received standard care

INTERVENTIONS:
Behavioral: PNMI — Eligible patients received patient navigator led plus mobile phone text messaging intervention (PNMI) or standard care. Bilingually trained patient navigators were recruited from our existing patient navigator training network, received intensive training on HBV prevention, diagnosis and treatment management, and served as a liaison with respective clinical partners. The PNMI intervention offered three education sessions on HBV management and weekly CHB patient-designed educational phone-based text messages for five weeks.
  Arms: behavioral PNMI

SUMMARY:
Asian Americans have the highest incidence, mortality and prevalence rates of hepatocellular carcinoma (HCC) among all U.S. racial and ethnic groups. The goal of this study is to investigate the efficacy of a Patient Navigator-led mobile phone text Messaging Intervention (PNMI) in improving hepatitis B follow-up care management for Asian Americans with chronic hepatitis B infection through a randomized controlled trial.

DETAILED DESCRIPTION:
Asian Americans have the highest incidence, mortality and prevalence rates of hepatocellular carcinoma (HCC) among all U.S. racial and ethnic groups. Inadequate chronic hepatitis B (CHB) monitoring and care are also likely to contribute to poorer outcomes and increased healthcare costs. The goal of this study is to investigate the efficacy of a Patient Navigator-led mobile phone text Messaging Intervention (PNMI) in improving hepatitis B follow-up care management for Asian Americans with chronic hepatitis B infection through a randomized controlled trial. The primary outcome of the study is Asian CHB patient adherence (measured as "having seen a doctor for CHB monitoring") to hepatitis B (HBV) monitoring guidelines at 6-month and 12-month assessments post-intervention.

Patient partners and stakeholders were engaged in all study stages. The findings of this study provided unique and promising opportunities for broadly disseminating and implementing the evidence-based intervention in the real-world practice, thus further preventing chronic liver diseases and reducing health disparities among high-risk underserved populations.

ELIGIBILITY:
Inclusion Criteria:

1. self-identified Chinese, Korean and Vietnamese ethnicity
2. age 18 and above
3. accessible by telephone with text message feature
4. presence in the same geographic study area for a period of one year
5. not enrolled in any chronic HBV adherence management intervention
6. medically diagnosed chronic HBV infection with positive for hepatitis B surface antigen (HBsAg) for more than six months, and
7. Never or non compliant with HBV monitoring guidelines.

Exclusion Criteria:

Patients were excluded from the study for the following conditions:

1. diagnosed with cirrhosis, hepatocellular carcinoma, liver failure and liver cancer
2. concurrent hepatitis C infection, and
3. concurrent HIV infection

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 532 (Actual)
Dates: Start 2014-09; Primary Completion 2018-01-31 (Actual); Study Completion 2018-01-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Grace X Ma, PhD, Principal Investigator — Temple University

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Ma GX, Zhu L, Tan Y, Zhai S, Ma X, Ogunwobi OO, Yang WJ, Ting T, Kim S, Wang MQ. A Comparative Trial of Improving Care for Underserved Asian Americans Infected with Hepatitis B Virus. Dig Dis Sci. 2023 Jun;68(6):2333-2343. doi: 10.1007/s10620-023-07840-5. Epub 2023 Feb 7. PMID 36749506

RESULTS

PARTICIPANT FLOW:
Groups:
- Behavioral PNMI: Eligible patients received patient navigator led plus mobile phone text messaging intervention (PNMI) or standard care. Bilingually trained patient navigators were recruited from our existing patient navigator training network, received intensive training on HBV prevention, diagnosis and treatment management, and served as a liaison with respective clinical partners. The PNMI intervention offered three education sessions on HBV management and weekly CHB patient-designed educational phone-based text messages for five weeks.
- Usual Care: eligible chronic HBV patients received usual care
Period: Overall Study Baseline
Arm/Group | Behavioral PNMI | Usual Care
Started | 272 | 260
Completed | 272 | 260
Not Completed | 0 | 0
Period: 6-month Follow-up
Arm/Group | Behavioral PNMI | Usual Care
Started | 272 | 260
Completed | 259 | 247
Not Completed | 13 | 13
Not completed — Lost to Follow-up | 8 | 7
Not completed — Withdrawal by Subject | 5 | 6
Period: 12-month Follow-up
Arm/Group | Behavioral PNMI | Usual Care
Started | 259 | 247
Completed | 248 | 231
Not Completed | 11 | 16
Not completed — Lost to Follow-up | 5 | 5
Not completed — Withdrawal by Subject | 6 | 11

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Behavioral PNMI | Usual Care | Total
Number analyzed (Participants) | 272 | 260 | 532
Age, Continuous [Mean (Full Range); unit: years] | 50 [20 to 88] | 49 [19 to 86] | 50 [19 to 88]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 119 | 133 | 252
  Male | 153 | 127 | 280
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Chinese | 225 | 216 | 441
  Vietnamese | 17 | 23 | 40
  Korean | 30 | 21 | 51
States of Residence [Count of Participants; unit: Participants]
  Pennsylvania/New Jersey | 164 | 160 | 324
  New York | 108 | 100 | 208

OUTCOME MEASURES:

1. Primary Outcome: Change of the Rates of Participants Who Adherent to Recommended Clinical Care for the Monitoring of Chronic HBV Infection
Description: The primary outcome is adherence to recommended clinical care for the monitoring of chronic HBV infection, specifically: 1) whether they visited doctors for their CHB, and 2) whether they received a blood test every 6 months such as alanine transaminase (ALT). All primary outcome measures were assessed at both the 6-month and 12-month follow-up surveys.
Time Frame: 6-month and 12-month follow up
Population: A total of 506 participants completed the 6-month follow-up assessment, among which 479 completed the 12-month follow-up assessment.
Measure: Count of Participants; unit: Participants
Arm/Group | Behavioral PNMI | Usual Care
Number analyzed (Participants) | 259 | 247
Participants
  Doctor's Visit by 6-month follow-up | 200 | 113
  Doctor's Visit by 12-month follow-up: number analyzed (Participants) | 248 | 231
  Doctor's Visit by 12-month follow-up | 225 | 140
  Blood Test (ALT) by 6-month follow-up | 137 | 62
  Blood Test (ALT) by 12-month follow-up: number analyzed (Participants) | 248 | 231
  Blood Test (ALT) by 12-month follow-up | 164 | 87

ADVERSE EVENTS:
Time Frame: through study completion, an average of 1 year
Arm/Group | Behavioral PNMI | Usual Care
All-Cause Mortality (participants affected / at risk) | 0/272 | 0/260
Serious Adverse Events (participants affected / at risk) | 0/272 | 0/260
Other Adverse Events (participants affected / at risk) | 0/272 | 0/260

LIMITATIONS AND CAVEATS:
In this study, we validated only those who reported their follow up visits and blood tests in collaboration with clinical partners; validating for all participants enrolled would be ideal. The results may not represent all Asian American groups.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2014-10-20): https://cdn.clinicaltrials.gov/large-docs/66/NCT02421666/Prot_SAP_000.pdf